CLINICAL TRIAL: NCT06017154
Title: The Acute Effects of Brain Activation and Functional Connectivity Following Motor-cognitive Training Using Functional MRI
Brief Title: Acute Effect of Motor-Cognitive Training
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ke'La H Porter (Other)
Responsible Party: Sponsor-Investigator, Ke'La H Porter, Research Analyst Principal, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 88851
Record Dates: First submitted 2023-08-18; First posted 2023-08-30 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Injury;Sports
Keywords: injury prevention; cognition; physical performance; athletic training
MeSH Terms: conditions — Athletic Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Physically active females (Experimental): Healthy active females between 18 and 25
  Interventions: Other: Motor-Cognitive Training Program

INTERVENTIONS:
Other: Motor-Cognitive Training Program — The training will incorporate cognitive tasks which focus on reaction time, processing speed, working memory, cognitive flexibility, and inhibitory control using visual stimuli on a screen or through sensors which illuminate using LED lights. These cognitive tasks will be performed while also executing physical performance tasks that challenge static and dynamic postural stability, lateral movement, agility, and other movement patterns. The training session will last approximately 30 minutes and participants will complete up to 5 exercises

SUMMARY:
Participants will complete a functional MRI to evaluate brain activation, functional connectivity, and behavioral performance immediately before and after a training program (approximately 30 minutes). The training program will comprise of integrate neuromuscular (agility, dynamic postural stability, shuffling, rapid acceleration/deceleration, plyometrics, lateral shuffle, and core stability) and cognitive (reaction time, processing speed, task switching, decision-making, and working memory) challenges.

ELIGIBILITY:
Inclusion Criteria:

* Physically active

Exclusion Criteria:

* Injury to the muscle or bone (upper extremity, lower extremity, or back) within the past 3 months
* Had musculoskeletal surgery or fracture (required open reduction internal fixation or within the last 12 months)
* Had a concussion or mild head injury within the last year
* Have been diagnosed with any kind of neurological, vestibular, or visual disturbance that impairs mobility
* Currently taking medications that affect the central nervous system
* Pregnant or suspicions of being pregnant
* Have metal fragments, pins, plates, or clips, shrapnel, body piercings that cannot be removed, have surgical implants or orthodontics that cannot be removed
* Have claustrophobia
* Have a history of cognitive impairment

Ages: 18 Years to 25 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 21 (Actual)
Dates: Start 2023-09-17 (Actual); Primary Completion 2024-02-05 (Actual); Study Completion 2024-02-05 (Actual)

PRIMARY OUTCOMES:
Change in brain activation | 2 hours, pre-training session and immediately post-training session
  During the task-based functional MRI scan the participant will complete a task-switching cognitive task, where participants have to identify two possible shapes (circle or square), in one of two possible colors (red or blue). They will respond using a trigger under their left and right foot. The level of brain activation during the task will be captured and reported.
Change in functional connectivity | 2 hours, pre-training session and immediately post-training session
  The participant will complete a resting-state functional MRI scan in which they will lay still in the scanner. No task is performed during this scan. Functional connectivity (functionally related regions of the brain that are co-activated) during the scan will be captured and reported.
Change in reaction time | 2 hours, pre-training session and immediately post-training session
  During the task-based functional MRI scan the participant will complete a task-switching cognitive task, where participants have to identify two possible shapes (circle or square), in one of two possible colors (red or blue). They will respond using a trigger under their left and right foot. The reaction time in milliseconds will be captured. The change in reaction time from pre to post training session will be reported.
Change in accuracy | 2 hours, pre-training session and immediately post-training session
  During the task-based functional MRI scan the participant will complete a task-switching cognitive task, where participants have to identify two possible shapes (circle or square), in one of two possible colors (red or blue). They will respond using a trigger under their left and right foot. The percent of correct responses (accuracy) will be captured. The change in accuracy from pre to post training session will be reported.

SECONDARY OUTCOMES:
Demographic/Injury History Form | Once, pre-training
  The demographic and injury history form is designed to capture: 1) information about the participant including age, height, weight, race, ethnicity, 2) information related to sports participation, and 3) information related to past injuries or medical conditions which are relevant to the study.
Defense Veterans Pain Rating Scale | Once, pre-training
  The Defense Veterans Pain Rating Scale is a valid 5-item scale to assess pain magnitude and pain interference. This scale ranges from 0 to 10, 0 indicating no pain/interference and 10 indicating as bas as it could be/complete interference.
Modified Disablement In Physically Active Scale | Once, pre-training
  16-item patient-reported outcome instrument that assesses physical and psychosocial status.This scale ranges from 0 to 4, 0 indicating no problem and 4 indicating severe.
NASA Physical Activity Survey | Once, pre-training
  This survey asks individuals to self-report their general physical activity over the past week. This survey ranges from 0 to 10, 0 indicating sedentary and 10 indicating high physical activity.
Heart rate | 35 minutes, during the training session
  Heart rate will be monitored with a noninvasive heart rate monitor that will be worn by the participant around the chest at the level of the xiphoid process. Resting heart rate will be collected prior to the start intervention then monitored and recorded throughout the training session.
Average reaction time during the intervention | 30 minutes, during the training session
  Average reaction time in milliseconds will be captured during the exercises via light sensors.
Misses during the training session | 30 minutes, during the training session
  The number of misses will be captured during the exercises via light sensors. A miss is considered when they deactivate the wrong sensor or don't deactivate the sensor quickly enough.
Hits during the training session | 30 minutes, during the training session
  The number of hits will be captured during the exercises via light sensors. A hit is considered when they deactivate the correct sensor.
Number of errors during the training session | 30 minutes, during the training session
  The number of errors will be captured during the exercises by visual observation. An error occurs when they do not complete they exercise correctly.
Rate of perceived exertion | 30 minutes, during the training session
  After each exercise the participant will be asked to rate their perceived exertion on a scale from 6 to 20, 6 indicating low perceived exertion and 20 indicating high perceived exertion
Perceived cognitive difficulty | 30 minutes, during the training session
  After each exercise the participant will be asked to rate their perceived cognitive difficulty on a scale from 1 to 10, 1 indicating low cognitive challenge and 10 indicating high cognitive challenge

CONTACTS AND LOCATIONS:
Overall Officials: Ke'La H Porter, MS, Principal Investigator — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No